CLINICAL TRIAL: NCT05047510
Title: An Evaluation Study of GPC3 Targeted Fluorescence Imaging to Guide the Surgery of Hepatocellular Carcinoma
Brief Title: GPC3 Targeted Fluorescence Image Guided Surgery of Hepatocellular Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Academy of Sciences (Other Government)
Responsible Party: Principal Investigator, Zeyu Zhang, PHD, Principal Investigator, Chinese Academy of Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Chinese Academy of Sciences
Record Dates: First submitted 2021-09-08; First posted 2021-09-17 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Anti-GPC3-IRDye800CW Intraoperative Fluorescence (Experimental): The patients will receive an injection of fluorophore (Anti-GPC3-IRDye800CW) before the surgery. Then intraoperative fluorescence imaging will be performed to guide lesion resection.
  Interventions: Drug: Anti-GPC3-IRDye800CW

INTERVENTIONS:
Drug: Anti-GPC3-IRDye800CW — Drug Injection: Anti-GPC3-IRDye800CW

SUMMARY:
This study is to evaluate whether intraoperative fluorescence imaging targeting GPC3 can aid improve the surgical accuracy of hepatocellular carcinoma.

The main purposes of this study include:

① To raise the detection rate of hepatocellular carcinoma intraoperatively using the novel NIR-II fluorescence molecular imaging and the GPC-3 targeted fluorophore.

② To validate the safety and effectiveness of the designed GPC-3 targeted fluorophore for clinical application.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have been diagnosed with hepatocellular carcinoma.
2. Planned to receive hepatectomy.
3. Liver function Child-Pugh A/B.
4. GPC-3 was validated highly expressed preoperatively.
5. Aged 18 to 75, and the expected lifetime is longer than 6 months.
6. Approved to sign the informed consent.

Exclusion Criteria:

1. Allergic to IRDye800.
2. Enrolled in other trials in the past 3 months.
3. Another malignant tumor was found.
4. Undesirable function of heart, lung, kidney, or any other organs.
5. Unable to tolerate a hepatectomy.
6. The researchers considered inappropriate to be included.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
HCC lesions | During hepatocellular resection surgery.
  Numbers of intraoperatively detected hepatocellular carcinoma lesions.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Zhuhai People's Hospital, Zhuhai, Guangdong
  - The Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan

IPD SHARING:
Plan to Share IPD: Undecided